CLINICAL TRIAL: NCT04294238
Title: Effects of Moderate Aerobic Exercise on the Proteome and Function Alteration of HDL Sub-Fractions in Male Youth With Abdominal Obesity
Brief Title: The Function and Proteome Alteration of HDL Subclass After Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingfeng Wang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SYSEC-KY-KS-2019-011
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: Obesity, Aerobic exercise, HDL subclass, Proteome, function
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Self-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-exercise (Experimental): The aerobic exercise intervention consisted of 12 weeks of aerobic exercise training of moderate intensity (about 75 percentage of peak heart rate) of 40-60 min per time, 3-5 times per week, at least 150 min per week.
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — The aerobic exercise intervention consisted of 12 weeks of aerobic exercise training of moderate intensity (about 75 percentage peak heart rate) of 40-60 min per time, 3-5 times per week, at least 150 min per week.

SUMMARY:
Obesity is one of the most important risk factors for cardiovascular disease (CVD). HDL protein composition can be altered without a change in cholesterol content. Alteration of the HDL proteome can result in dysfunctional HDL particles with reduced ability to protect against CVD. The aim of this study was to evaluate the influence of moderate aerobic exercise on HDL protein composition and its related function. This was a self-control study including 6 inactive male youths with abdominal obesity. HDL functions and its associations with proteome alteration would be analysized.

DETAILED DESCRIPTION:
The aim of present study is to test the effects of 12-week moderate aerobic exercise on the proteome and function alteration of HDL sub-fractions in male youth with abdominal obesity.

Study participants: youth males with abdominal obesity between the ages of 18 and 30 years were eligible for participation. Exclusion criteria were cardiovascular disease, diabetes or other chronic diseases, treatment with any medications, and had surgical procedures within the last 6 months. This study was approved by the Medical Ethics Committee at the Sun Yat-sen Memorial Hospital, complies with the Declaration of Helsinki principles and written informed consent would be obtained from all participants.

Data collection: anthropometric measurements, physical examination and blood samples were collected at 0 and 12 weeks. Cardiorespiratory measurements of each participant was measured using a bicycle-based graded exercise test at baseline.

Intervention: the exercise intervention consisted of 12 weeks of aerobic exercise training of moderate intensity (about 75 percentage of peak heart rate) of 40-60 min per time, 3-5 times per week, at least 150 min per week. All participants were instructed to maintain their usual dietary intakes. Completing a minimum of 80 percentage training sessions was satisfactory.

HDL isolation: HDL particles were fractionated into small, medium and large (S/M/L)-HDL subfractions by an ÄKTA fast protein liquid chromatography (FPLC) system.

Proteomics Experiments: equal volumes of L/M/S-HDL subclass were applied to the CSH resin, trypsinized, and then recognized via LC-MS. HDL proteins in HDL subclass were detected by MS-based label-free quantitation

HDL functions: cholesterol efflux capacity, anti-inflammation and anti-oxidative capacity, endothelial protective function

Analysis: data are expressed as mean and SD for continuous variables, or percentage for category variables. Difference of variables between baseline and after exercise were compared using analysis of Paired t-test or Mann Whitney U test. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inactive youth males with abdominal obesity: BMI>28 (weight in kilograms divided by height in meters squared) and weight stable for 6 months, waist to height ratio was ≥0.5 and/or waist circumference was ≥102 centimetres between the ages of 18 and 30 years.

Exclusion Criteria:

* Participants with cardiovascular disease, diabetes or other chronic diseases, treatment with any medications, and had surgical procedures within the last 6 months.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The percentage change of HDL cholesterol efflux capacity | 12 week
  The primary outcome was the mearsurement of HDL function for removing excess cholesterol from peripheral cells
Proteome alteration of HDL subclass | 12 week
  HDL proteome was analyzed by mass spectrometry using label-free protein quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfeng Wang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Due to restrictions that protect participant privacy, data are available upon request. The data ( study protocol) will be available upon request to all interested researchers.
Supporting Information: Study Protocol
Time Frame: The data will become available at 01/01/2021 and for 1 year.